CLINICAL TRIAL: NCT03949114
Title: Early Rehabilitation Intervention on Prevention of Postoperative Delirium in Neurosurgical Patients
Brief Title: Rehabilitation Intervention on Prevention of Postoperative Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, zhuminglan, nurse manger, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-022
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Delirium; Eras
Keywords: neurosurgery
MeSH Terms: conditions — Delirium | interventions — Nursing Care; Rehabilitation

STUDY DESIGN:
Intervention Model Description: During the period from June 1, 2019 to December 31, 2019, 150 patients with craniotomy who met the criteria and signed informed consent were included in the control group, from January 1, 2020 to June 30, 2020. During the period, 150 patients who met the standard neurosurgical craniotomy were included in the observation group.
Who Masked: Outcomes Assessor
Masking Description: Responsible nurses will conduct daily life skills and sputum assessments for all patients, and the data collector will collect the data needed for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): 1) Performing a weak debilitating phenotype screening on the patients before surgery;
  (2) Do the early rehabilitation intervention process:
  Interventions: Behavioral: Evaluation; Behavioral: rehabilitation
- Control group (Active Comparator): 1) Performing a weak debilitating phenotype screening on the patients before surgery; (2) Patients in the control group were treated according to the general nursing routine after neurosurgery;
  Interventions: Behavioral: Evaluation; Behavioral: nursing care

INTERVENTIONS:
Behavioral: Evaluation — Evaluate a weak debilitating phenotype screening on the patients before surgery;
  Other Names: Fried assessment
Behavioral: nursing care — Traditional post-operative nursing care
  Other Names: post-operative nursing care
  Arms: Control group
Behavioral: rehabilitation — 1. Postoperative vital signs were stabilized for 2 hours and then assisted to turn over; 2 to 3 hours to change position, awake without swallowing dysfunction, to fluid diet; 6 hours later, raise the bed 15 to 30 °, eat a half-flow diet.
  2. On the first day after surgery, raise the bed 45 °, row and position training; catheter clamping training; assessment of pain, preventive analgesia. Early rehabilitation training was performed for 60 minutes each time for 5 consecutive days.
  Other Names: ERAS
  Arms: test group

SUMMARY:
1. A questionnaire on "Cognition and Attitudes of Nurses on Postoperative Deafness in Neurosurgical Patients" was initially formed through reference literature and expert opinions. The content includes two dimensions of knowledge and attitude, all of which are single-choice questions. There are 11 items in the knowledge dimension, 1 point for the correct answer, 0 point for the wrong answer, and 0 to 11 points for the total score. The average score is the average score and the score of the score is the average score. The average score is ≤60%. Knowledge; attitude dimension is 7 items, using the Likert 4 rating method, "very disagree ~ very agree" count "1 to 4 points", total score 7 to 28 points. A sample questionnaire survey was conducted among non-severe unit nurses in the top three hospitals in the province to understand the level of cognitive mastery of the neurosurgical nurses in the province and the current status of interventions, and to compare the attitudes of nurses with different academic qualifications, years of work and work experience to postoperative intervention. And the level of knowledge mastery.
2. Patients who underwent surgery on the neurosurgery in our hospital from December 31, 2010 to December 31, 2019 were used as the control group. After informed notification, the patients with the enrollment conditions were screened for Fried's debilitating phenotype and performed. Post-routine care; patients who underwent craniotomy in our department of neurosurgery from January 1, 2020 to June 31, 2020 were included in the intervention. Patients who met the criteria for admission were informed and informed consent was obtained. Develop an early rehabilitation process to guide patients to systematic early rehabilitation training. To compare the incidence of debilitating, sputum incidence (Nursing Delirium Screening Scale, Nu-DESC), sputum-related adverse events, Activity of Daily Living (ADL), patient satisfaction, etc. The clinical application effect of the early rehabilitation intervention system.

DETAILED DESCRIPTION:
Research method: This project includes two parts of research.

Study 1:

1.1 Research object 1.1.1 Research population: 5 nurses in the top three hospitals in Zhejiang Province Exclusions: training nurses, rotation nurses, and nurses who have been working for <1 year.

1.1.2 Sample size: 80 people 1.2 Time: January 2019 - June 2019 1.3 Content

1. Through self-designed questionnaires (see Attachment 1), the questionnaires cover the general information of the respondents including gender, age, working years, professional titles, academic qualifications, etc., including basic knowledge of postoperative sputum, and current preventive measures , knowledge needs and other aspects. The questionnaires on postoperative delirium knowledge were divided into two parts: subjective and objective. It mainly includes the concept of postoperative delirium, clinical manifestations, contents of nurses' evaluation form, diagnosis and treatment, risk factors and hazards. For the subjective and objective knowledge points, the choice is the main form.
2. The questionnaire was distributed on the spot to 80 nurses in the top three hospitals in Zhejiang Province. The knowledge dimension consisted of 11 items. The correct answer was 1 point, the wrong score was 0 points, and the total score was 0 to 11 points. The percentage of points and full marks is taken as the average scoring rate. The average scoring rate is ≤60%, which means that the nurses fail to master the relevant knowledge; the attitude dimension is 7 items, and the Likert 4 level is used. "Very disagree~very agree" ~4 points", the total score is 7 to 28 points. The important information can not be filled out as a complete questionnaire.
3. According to the working years of less than 3 years, 4 to 10 years, more than 10 years, the nursing staff can be divided into three levels: low, medium and high. The level of knowledge and attitude of the nursing staff at different levels are compared.

1.4 Method: Statistical analysis was performed using SPSS 22.0 software. The measurement data that conforms to the normal distribution is described by the mean value and the standard deviation, and the measurement data that does not conform to the normal distribution are described by the median and the interquartile range. The count data is described by a pie chart or a bar chart. In the stratified analysis, the comparison of the measurement data that conforms to the normal and the homogeneity of the variance is performed by t test or ANOVA. The comparison of the measurement data that does not conform to the normality or the homogeneity of the variance is performed by nonparametric test, and the comparison of the count data is performed by chi-square test. .

Study 2:

2.1. Research object 2.1.1 Study population: patients after neurosurgery 2.1.2 Research time: 2011.06-2020.06 2.1.3 Sample size: 300 people; 2.1.4 Inclusion criteria:

1. Age ≥ 18 years old, <75 years old, gender is not limited;
2. Those with clear consciousness after neurosurgery craniotomy;
3. Sign the research informed consent form. 2.1.4 Exclusion criteria:

1) The patient has a history of cognitive dysfunction, mental illness, senile dementia, and stroke before surgery; 2) Patients and their families with poor behavioral compliance; 3) Patients with drug dependence and alcohol dependence; 4) Serious postoperative complications (such as infection, bleeding, etc.). 2.1.5 Elimination criteria:

1) Patients who have changed their condition during the study, or who have been transferred, discharged, and died.

2.2 Grouping method: During the period from June 1, 2019 to December 31, 2019, 150 patients with craniotomy who met the criteria and signed informed consent were included in the control group, from January 1, 2020 to June 30, 2020. During the period, 150 patients who met the standard neurosurgical craniotomy were included in the observation group.

2.3 Content:

(1) Performing a weak debilitating phenotype screening on the patients before surgery; (2) Patients in the control group were treated according to the general nursing routine after neurosurgery; (2) The observation group implements the early rehabilitation intervention process:

1. Postoperative vital signs were stabilized for 2 hours and then assisted to turn over; 2 to 3 hours to change position, awake without swallowing dysfunction, to fluid diet; 6 hours later, raise the bed 15 to 30 °, eat a half-flow diet.
2. On the first day after surgery, raise the bed 45 °, row and position training; catheter clamping training; assessment of pain, preventive analgesia. Early rehabilitation training was performed for 60 minutes each time for 5 consecutive days. The details are as follows:

   1. Active or passive assisted state of extension of the shoulder, elbow, ankle and knee joints to maximize the extent of movement of the distal extremity to prevent contracture. (10 minutes).
   2. Strength training (10 minutes) for the trunk and upper and lower limbs under active or passive assistance.
   3. Strengthen the functional training of the upper limbs and hand fine movements (15 minutes).
   4. Balance training, starting with the sitting position and gradually transitioning to the station position, especially after the patient can complete the standing movement (even in the case of assistance), strengthen the training of standing balance (10 minutes).
   5. Walk back and forth with assistance and gradually transition to walking back and forth (15 minutes) with only surveillance protection.
3. From the second day after surgery to five days after surgery, daily daily life training, including washing, dressing, eating, etc. Walk 2 times a day for 30 minutes each time.
4. The rest of the care is the same as general postoperative care routine. (4) Urgent treatment, once the patient is found to have timely treatment intervention, including drug and non-drug treatment.

2.4 Observation indicators and observation time 2.4.1 Observation time

1. T1: return to the ward after surgery to 5 days after surgery;
2. T2: at the time of discharge;
3. T3: 1 week after discharge;
4. T4: 1 month after discharge. 2.4.2 Observation indicators

(1) T: Phase 1 MAIN OUTCOME MEASURES: Debilitating index, incidence of delirium. Secondary observation indicators: 谵妄 related adverse events (accident extubation, falls, etc.); (2) T2 phase: Postoperative hospital stay, hospitalization expenses, and activities of daily living activities, using the Barthel Index (BI), patient satisfaction (3) T3: the ability of daily living activities; (4) T4: activities of daily living activities

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clear consciousness after neurosurgery craniotomy;
2. Sign the research informed consent form.

Exclusion Criteria:

1. Patients have a history of cognitive dysfunction, mental illness, senile dementia, and stroke before surgery;
2. Patients and their families with poor behavioral compliance;
3. Patients with drug dependence and alcohol dependence; -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of postoperative delirium | The first to fifth day after surgery
  use the NU-DESC to assess every postoperative patients,to see the incidence of postoperative delirium

OTHER OUTCOMES:
Daily life ability | One week after discharged
  Use Barthel Index to assess the activity of daily living ability
Daily life ability | One month after discharged
  Use Barthel Index to assess the activity of daily living ability

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes